CLINICAL TRIAL: NCT01591096
Title: Thrombolysis in Pediatric Stroke (TIPS)
Acronym: TIPS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of patient accrual
Sponsor: Seattle Children's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other); Medical College of Wisconsin (Other); University of Texas at Austin (Other); Alberta Children's Hospital (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Catherine Amlie-Lefond, Associate Professor of Neurology, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01NS065818 (NIH)
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Stroke
Keywords: Stroke; Childhood; Thrombolysis
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tissue plasminogen activator (Experimental): All patients will receive study drug.
  Interventions: Drug: Tissue plasminogen activator (Activase®)

INTERVENTIONS:
Drug: Tissue plasminogen activator (Activase®) — Investigation labeled tPA will be obtained for all sites by the Core Pharmacy as commercially available recombinant tPA (Genentech as Activase®) for IV administration. The Bayesian method of toxicity probability intervals will be used to select one of the following three dose tiers (0.75, 0.9, 1.0 mg/kg) of IV tPA. The dose escalation for the two age groups (2-10, 11-17 years) will be performed independently. The maximum dose for each tier will be reached at a weight of 90 kg.
  Other Names: Genentech as Activase®

SUMMARY:
Thrombolysis in Pediatric Stroke (TIPS) is a five-year multi-center international safety and dose-finding study of intravenous (IV) tPA in children with acute ischemic stroke (AIS) to determine the maximal safe dose of intravenous Tissue Plasminogen Activator (IV-tPA) among three doses (0.75. 0.9, 1.0 mg/kg) for children age 2-17 years within 4.5 hours from onset of acute AIS.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To determine the maximal safe dose of intravenous (IV) tPA among three doses (0.75. 0.9, 1.0 mg/kg) for children age 2-17 years within 4.5 hours from onset of acute AIS.
2. To determine the pharmacokinetics of tPA and its inhibitor, plasminogen activator inhibitor in these children.
3. To measure the 3-month neurological outcome in children treated with IV tPA.

TRIAL DESIGN:

Thrombolysis in Pediatric Stroke (TIPS) is a five-year multi-center international safety and dose-finding study of intravenous (IV) tPA in children with acute AIS to determine the maximal safe dose of intravenous (IV) tPA among three doses (0.75. 0.9, 1.0 mg/kg) for children age 2-17 years within 4.5 hours from onset of acute AIS.

An adaptive dose finding method will be applied to escalate across the three dose levels within two age groups: 2-10 years (prepubertal) and 11-17 years. Dose will be escalated based on safety (absence of excess toxicity) with at least 3 children treated at each dose level. Intracranial hemorrhage following stroke can occur even in the absence of thrombolytic therapy, but the risk is increased by the use of thrombolytics.

Primary endpoint toxicity is defined as SICH or severe hemorrhage within 36 hours of tPA administration, defined as any of the following:

1. PH2 (parenchymal hemorrhage within 36 hours after tPA administration involving > 30% of the infarcted area), regardless of whether or not it is associated with clinical deterioration, OR,
2. Any intracranial hemorrhage which is judged to be the most important cause of neurological deterioration. Neurological deterioration is guided by a minimum of change of 2 or more points on the PedNIHSS from the lowest PedNIHSS. At the time of each PedNIHSS assessment, the site PI or co-PI will review the patient's course with the care team to ensure that all changes in neurologic status, including improvements since the last assessment by the study team, are captured, OR,
3. Any hemorrhage that results in the need for transfusion, need to discontinue study drug, surgical evacuation of hemorrhage, or death.

TIPS will determine the pharmacokinetics of tPA and its inhibitor, plasminogen activator inhibitor, including free tPA, PAI-1, and tPA antigen in children receiving IV tPA for acute AIS. In addition, TIPS will measure the 3-month neurological outcome in children treated with IV tPA.

TRIAL POPULATION:

TIPS will enroll a maximum of 18 children age 2-10 years and maximum of 18 children age 11-17 years within 4.5 hours of the onset of acute AIS. On MRA or CTA they will have partial or complete occlusion of the artery, consistent with focal impairment of the arterial flow, that correlates with the clinical deficit.

TIPS STUDY INTERVENTION:

Investigation labeled tPA will be obtained for all sites by the Core Pharmacy as commercially available recombinant tPA (Genentech as Activase®) for IV administration. The Bayesian method of toxicity probability intervals will be used to select one of the following three dose tiers (0.75, 0.9, 1.0 mg/kg) of IV tPA. The dose escalation for the two age groups (2-10, 11-17 years) will be performed independently. The maximum dose for each tier will be reached at a weight of 90 kg.

ELIGIBILITY:
To be eligible for TIPS, a patient must meet the following Inclusion Criteria:

1. Age 2 to 17 years inclusive.
2. Clinical presentation consisting of clearly defined acute onset of neurological deficit in a pattern consistent with arterial territory ischemia.
3. Clinically significant deficit as defined by a PedNIHSS score of ≥ 6 and ≤ 24 felt to be due to acute stroke that is not improving at the time of initiation of tPA administration
4. Time of symptom onset within 4.5 hours of initiation of treatment for IV tPA. Time of symptom onset is defined as time the patient was last seen awake and at neurological baseline.
5. Radiological confirmation of an acute arterial ischemic stroke in one of two ways:

   * MRI confirmation, consisting of acute infarction with restricted diffusion in an arterial territory consistent with the clinical syndrome plus MRA showing partial or complete occlusion in an intracranial artery corresponding to the infarct location, OR,
   * CT and CT angiogram confirmation, consisting of normal head CT or early hypodensity in an arterial territory consistent with the clinical syndrome plus CT angiogram showing partial or complete occlusion in an intracranial artery corresponding to the infarct location.
6. Baseline neuroimaging (CT or MRI) with no evidence of intracranial hemorrhage (including HI-1, HI-2, PH-1 or PH-2). If no head CT scan is done, the pre-tPA MRI must include Gradient-recalled ECHO (GRE) imaging or Susceptibility Weighted Imaging (SWI) sequences.
7. Children with seizures at or following onset of stroke may be included, as long as the clinical picture is consistent with the documented arterial occlusion.

3.4.1.2.2. Patients with the following Exclusion Criteria will not be eligible for TIPS:

Safety Related exclusion criteria:

1. Patients in whom time of symptom onset is unknown.
2. Pregnancy
3. Clinical presentation suggestive of subarachnoid hemorrhage (SAH), even if head CT or head MRI scan is negative for blood.
4. Patient who would decline blood transfusion if indicated
5. History of prior intracranial hemorrhage
6. Known cerebral arterial venous malformation, aneurysm, or neoplasm
7. Persistent Systolic Blood Pressure > 15% above the 95th percentile for age while sitting or supine
8. Glucose < 50 mg/dl (2.78 mmol/l) or > 400 mg/dl (22.22 mmol/l)
9. Bleeding diathesis including platelets < 100,000, PT > 15 sec (INR > 1.4) or elevated PTT > upper limits of the normal range.
10. Clinical presentation consistent with acute myocardial infarction (MI) or post-MI pericarditis that requires evaluation by cardiology prior to treatment
11. Stroke, major head trauma, or intracranial surgery within the past 3 months
12. Major surgery or parenchymal biopsy within 10 days (relative contraindication)
13. Gastrointestinal or urinary bleeding within 21 days (relative contraindication)
14. Arterial puncture at noncompressible site or lumbar puncture within 7 days (relative contraindication). Patients who have had a cardiac catheterization via a compressible artery are not excluded.
15. Patient with malignancy or within 1 month of completion of treatment for cancer
16. Patients with an underlying significant bleeding disorder. Patients with a mild platelet dysfunction, mild von Willebrand Disease or other mild bleeding disorders are not excluded.

Stroke related exclusions:

1. Mild deficit (PedNIHSS < 6) at start of tPA infusion
2. Severe deficit suggesting very large territory stroke, with pre-tPA PedNIHSS > 25, regardless of the infarct volume seen on neuroimaging
3. Stroke suspected to be due to subacute bacterial endocarditis, moyamoya, sickle cell disease, meningitis, bone marrow, air or fat embolism
4. Previously diagnosed primary angiitis of the central nervous system (PACNS) or secondary CNS vasculitis. Focal cerebral arteriopathy (FCA) of childhood is not a contraindication.

Neuro-imaging related exclusions:

1. Intracranial hemorrhage (HI-1, HI-2, PH-1 or PH-2) on pretreatment head MRI or head CT
2. Intracranial dissection (defined as at or distal to the opthalmic artery)
3. Large infarct volume, defined by the finding of acute infarct on MRI involving 1/3 or or more of the complete MCA territory involvement, regardless of the pre-tPA PedNIHSS score due to increased risk of ICH.78, 79

Drug Related exclusions:

1. Known allergy to recombinant tissue plasminogen activator
2. Patient on anticoagulation therapy must have INR ≤ 1.4
3. Patient who received heparin within 4 hours must have aPTT in normal range
4. LMWH within past 24 hours (aPTT and INR will not reflect LMWH effect)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Amlie-Lefond, MD, Principal Investigator — Seattle Children's Hospital
Locations (15):
- United States (13):
  - Stanford University and Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center at Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Medical School at Houston, Houston, Texas
  - The University of Utah and Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rivkin MJ, deVeber G, Ichord RN, Kirton A, Chan AK, Hovinga CA, Gill JC, Szabo A, Hill MD, Scholz K, Amlie-Lefond C. Thrombolysis in pediatric stroke study. Stroke. 2015 Mar;46(3):880-5. doi: 10.1161/STROKEAHA.114.008210. Epub 2015 Jan 22. No abstract available. PMID 25613306
- [Result] Bernard TJ, Rivkin MJ, Scholz K, deVeber G, Kirton A, Gill JC, Chan AK, Hovinga CA, Ichord RN, Grotta JC, Jordan LC, Benedict S, Friedman NR, Dowling MM, Elbers J, Torres M, Sultan S, Cummings DD, Grabowski EF, McMillan HJ, Beslow LA, Amlie-Lefond C; Thrombolysis in Pediatric Stroke Study. Emergence of the primary pediatric stroke center: impact of the thrombolysis in pediatric stroke trial. Stroke. 2014 Jul;45(7):2018-23. doi: 10.1161/STROKEAHA.114.004919. Epub 2014 Jun 10. PMID 24916908

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was recruited for the study, however, they did not receive the intervention due to an AE
Period: Overall Study
Arm/Group | Tissue Plasminogen Activator
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tissue Plasminogen Activator
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Intracranial Hemorrhage
Description: Any PH 2 OR, Any intracranial hemorrhage which is judged to be the most important cause of neurological deterioration (a minimum of change of 2 or more points on the PedNIHSS from the lowest PedNIHSS). At the time of each PedNIHSS assessment, the site PI or co-PI will review the patient's course with the care team to ensure that all changes in neurologic status, including improvements since the last assessment by the study team, are captured, OR, Any hemorrhage that results in the need for transfusion, need to discontinue study drug, surgical evacuation of hemorrhage, or death.
Time Frame: 36 hours
Population: Data cannot be reported in the data table as no data was collected
Arm/Group | Tissue Plasminogen Activator
Number analyzed (Participants) | 0

2. Secondary Outcome: Pharmacokinetics of tPA
Description: TIPS will determine the pharmacokinetics of tPA and its inhibitor, plasminogen activator inhibitor, including free tPA, PAI-1, and tPA antigen in children receiving IV tPA for acute AIS. In addition, TIPS will measure the 3-month neurological outcome in children treated with IV tPA.
Time Frame: 24 hours
Population: Data cannot be reported in the data table as no data was collected
Arm/Group | Tissue Plasminogen Activator
Number analyzed (Participants) | 0

3. Secondary Outcome: Pharmacokinetics of tPA
Description: as for outcome 2
Time Frame: 24 hours
Population: Data cannot be reported in the data table as no data was collected
Arm/Group | Tissue Plasminogen Activator
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Tissue Plasminogen Activator
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Tissue Plasminogen Activator
Hypoventilation, bradycardia (Cardiac disorders) | 1/1 (1) — Patient developed hypoventilation and bradycardia after extubation following sedation for head MRI and MRA. (no tPA given).

LIMITATIONS AND CAVEATS:
Early termination due to lack of participant accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No